CLINICAL TRIAL: NCT06888362
Title: A Double-blind, Randomised, Placebo-controlled Phase I Trial to Investigate Safety, Tolerability and Pharmacokinetics of Single Ascending Topical Doses of GZ21T in Healthy Volunteers
Brief Title: Trial to Investigate GZ21T in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzada Pharmaceuticals USA, Inc. (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: A24-0001..; 2024-512893-86-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-15; First posted 2025-03-21 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Part A:
  * Cohort 1: 25.5 mg/cm2 GZ21T or placebo will be applied to 900 cm2 of the skin, corresponding to approximately 5% body surface area (BSA) and 23 g cream.
  * Cohort 2: 25.5 mg/cm2 GZ21T or placebo will be applied to 1350 cm2 of the skin, corresponding to approximately 7.5% BSA and 35 g cream.
  * Cohort 3: 25.5 mg/cm2 GZ21T or placebo will be applied to 1800 cm2 of the skin, corresponding to approximately 10% BSA and 46 g cream.
  * Cohort 4: 25.5 mg/cm2 GZ21T or placebo will be applied to the face, corresponding to approximately 3-3.5% BSA (540 - 630% cm2) and 16 g cream.
  Part B:
  * Cohort 1: 13 mg/cm2 GZ21T will be applied to 900 cm2 of the skin, corresponding to approximately 5% body surface area (BSA)
  * Optional cohorts 2 and 3: A single dose of GZ21T decided based on the results from preceding cohorts will be applied to 900 cm2 of the skin corresponding to approximately 5% BSA.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A: Double-blind Part B: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A, Cohort 1 (Experimental): 25.5 mg/cm2 GZ21T or placebo will be applied to 900 cm2 of the skin, corresponding to approximately 5% body surface area (BSA) and 23 g cream.
  Interventions: Drug: GZ21T
- Part A, Cohort 2 (Experimental): 25.5 mg/cm2 GZ21T or placebo will be applied to 1350 cm2 of the skin, corresponding to approximately 7.5% BSA and 35 g cream.
  Interventions: Drug: GZ21T
- Part A, Cohort 3 (Experimental): 25.5 mg/cm2 GZ21T or placebo will be applied to 1800 cm2 of the skin, corresponding to approximately 10% BSA and 46 g cream.
  Interventions: Drug: GZ21T
- Part A, Cohort 4: (Experimental): 25.5 mg/cm2 GZ21T or placebo will be applied to the face, corresponding to approximately 3-3.5% BSA (540 - 630% cm2) and 16 g cream.
  Interventions: Drug: GZ21T
- Part B, Cohort 1 (Experimental): 13 mg/cm2 GZ21T will be applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 11.7 g cream
  Interventions: Drug: GZ21T
- Part B, Cohort 2 (Experimental): A single dose of GZ21T decided based on the results from preceding cohorts will be applied to 900 cm2 of the skin, corresponding to approximately 5% BSA
  Interventions: Drug: GZ21T
- Part B, Cohort 3 (Experimental): A single dose of GZ21T decided based on the results from preceding cohorts will be applied to 900 cm2 of the skin, corresponding to approximately 5% BSA
  Interventions: Drug: GZ21T

INTERVENTIONS:
Drug: GZ21T — GZ21T cream is intended to be studied as a potential treatment for patients with actinic keratoses and other dermatologic conditions which may be amendable to the study treatment.

SUMMARY:
This is a double-blind, randomised, placebo-controlled trial designed to evaluate safety, tolerability, and pharmacokinetics (PK) after topical administration of single ascending doses of GZ21T in healthy volunteers.

DETAILED DESCRIPTION:
Participants will receive a single topical application of GZ21T or placebo:

Part A:

* Cohort 1: 25.5 mg/cm2 GZ21T or placebo will be applied to 900 cm2 of the skin, corresponding to approximately 5% body surface area (BSA) and 23 g cream.
* Cohort 2: 25.5 mg/cm2 GZ21T or placebo will be applied to 1350 cm2 of the skin, corresponding to approximately 7.5% BSA and 35 g cream.
* Cohort 3: 25.5 mg/cm2 GZ21T or placebo will be applied to 1800 cm2 of the skin, corresponding to approximately 10% BSA and 46 g cream.
* Cohort 4: 25.5 mg/cm2 GZ21T or placebo will be applied to the face, corresponding to approximately 3-3.5% BSA (540 - 630% cm2) and 16 g cream.

Participants will come for 3 visits to the research clinic for screening, treatment, and follow-up.

Sentinel dosing will be applied. All participants will be carefully monitored by clinical staff during and after IMP application and will remain at the research clinic for at least 24 hours after treatment (Day 2) for safety assessments, including safety laboratory testing, 12-lead ECG, vital signs, local tolerability, physical examination and AEs, and PK assessments.

Part B:

* Cohort 1: 13 mg/cm2 GZ21T will be applied to 900 cm2 of the skin, corresponding to approximately 5% body surface area (BSA)
* Optional cohorts 2 and 3: A single dose of GZ21T decided based on the results from preceding cohorts will be applied to 900 cm2 of the skin corresponding to approximately 5% BSA. Participants will come for 3 visits to the research clinic and 1 telephone visit for screening, treatment, and follow-up.

All participants will be carefully monitored by clinical staff during and after IMP application and will remain at the research clinic for 2 hours after treatment for local tolerability and AE evaluation. On Day 2 (Visit 3), approximately 24 hours post-dose, participants will visit the research clinic for follow-up of local tolerability and AEs. A remote telephone call will be performed on Day 7 (Visit 4) to follow-up on local tolerability and AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial.
2. Healthy male or female participant aged 18 to 70 years, inclusive.
3. Body Mass Index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 at the time of the screening visit.
4. WOCBP must practice abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) or must agree to use a highly effective method of contraception with a failure rate of <1 % to prevent pregnancy from at least 2 weeks prior to the administration of IMP to 4 weeks after the last administration of IMP. In addition, any male partner of a female participant must, unless he is sterile (e.g., has undergone vasectomy), agree to use a condom from the first administration of IMP until 4 weeks after the last administration of IMP.

WOCBP must refrain from donating eggs from the first IMP administration until 3 months after the last IMP administration.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial or influence the results or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of IMP.
3. Any clinically significant abnormalities regarding physical examination, vital signs, 12- lead ECG, and laboratory values at the time of the screening visit, as judged by the Investigator.
4. Malignancy within the past 5 years, including removal of basal cell carcinoma.
5. Any planned major surgery within the duration of the trial.
6. Any skin condition including tattoos that may limit the evaluation of e.g., local tolerability as judged by the Investigator.
7. History of chronic urticaria, known history of urticaria triggered by specific factors or currently experiencing an episode of urticaria within the past 3 months.
8. History of psoriasis, atopic eczema and similar conditions, as judged by the Investigator.
9. Prescence of body hair or tattoos on the intended application areas, which in the opinion of the Investigator could interfere with local tolerability assessments.
10. Females who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
11. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis B and C antibodies and/or human immunodeficiency virus (HIV).
12. After 10 minutes of supine rest at the screening visit, any vital signs values outside the following ranges: - Systolic blood pressure: <90 or ≥140 mmHg, or - Diastolic blood pressure <50 or ≥90 mmHg, or - Pulse <40 or >90 bpm
13. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the screening visit, as judged by the Investigator.
14. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs or food with a similar chemical structure or class to GZ21T.
15. Regular use of any prescribed or non-prescribed medications, including antacids, analgesics, herbal remedies, within 2 weeks prior to the (first) administration of IMP, except occasional intake of paracetamol (maximum 2000 mg/day and not exceeding 3000 mg/week), as well as nasal decongestants without cortisone, antihistamine, or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
16. Unwillingness to abstain from the use of topical treatment (including but not limited to corticosteroids, calcineurin inhibitors, vitamin D analogues, and retinoids) at the application site within 1 week prior to Day 1 and from the use of moisturising ointment cream, emollients, oils (including shower oil) or sunscreen within 24 hours prior to Day 1 until 1 week after IMP administration.
17. Planned treatment or treatment with another investigational drug within 3 months prior to Day 1. Participants who consented and screened but were not dosed in previous clinical trials are not to be excluded.
18. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times per week is allowed before screening visit.
19. Positive screening result for drugs of abuse or alcohol at the screening visit or on admission to the trial site prior to the administration of the IMP. (Positive results that are expected given the participant's medical history and prescribed medications can be disregarded as judged by the Investigator.)
20. History of alcohol abuse or excessive intake of alcohol, history or presence of drug abuse including anabolic steroids, as judged by the Investigator.
21. Plasma donation within approximately 1 month of screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening, at the discretion of the Investigator.
22. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron West, Study Director — Ankh Life Sciences Limited
Locations (1):
- CTC (Clinical Trial Consultants) AB, Uppsala, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Cohort 1: 25.5 mg/cm2 GZ21T was applied to 900 cm2 of the skin, corresponding to approximately 5% body surface area (BSA) and 23 g cream.
- Part A, Cohort 2: 25.5 mg/cm2 GZ21T was applied to 1350 cm2 of the skin, corresponding to approximately 7.5% BSA and 35 g cream.
- Part A, Cohort 3: 25.5 mg/cm2 GZ21T was applied to 1800 cm2 of the skin, corresponding to approximately 10% BSA and 46 g cream.
- Part A, Cohort 4: 25.5 mg/cm2 GZ21T was applied to the face, corresponding to approximately 3-3.5% BSA and 16 g cream.
- Part A: Placebo: Corresponding amount of placebo was applied to the corresponding treatment area as the active treatment in Cohorts 1-4 in Part A.
- Part B, Cohort 1: 13 mg/cm2 GZ21T was applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 12 g cream.
- Part B, Cohort 2: 8 mg/cm2 GZ21T was applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 7 g cream.
- Part B, Cohort 3: 6,5 mg/cm2 GZ21T was applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 6 g cream.
Period: Overall Study
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo | Part B, Cohort 1 | Part B, Cohort 2 | Part B, Cohort 3
Started | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3
Completed | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo | Part B, Cohort 1 | Part B, Cohort 2 | Part B, Cohort 3 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 5 | 6 | 8 | 2 | 3 | 3 | 35
  >=65 years | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (16.6) | 62.2 (5.8) | 47.0 (21.6) | 39.7 (9.9) | 39.5 (17.8) | 25.0 (2.6) | 20.3 (1.2) | 37.3 (27.5) | 40.7 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 3 | 30
  Male | 3 | 3 | 3 | 0 | 2 | 0 | 0 | 0 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 8 | 3 | 2 | 3 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3 | 41

OUTCOME MEASURES:

1. Primary Outcome: AE
Description: Number of reported adverse events (AEs).
Time Frame: Day 1 to Day 7
Population: Full analysis set (FAS) consisted of all enrolled participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo | Part B, Cohort 1 | Part B, Cohort 2 | Part B, Cohort 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3
participants
  Any AE | 3 | 0 | 2 | 3 | 3 | 1 | 1 | 0
  Any SAE | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Causality: not related | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
  Causality: unlikely related | 3 | 0 | 1 | 2 | 2 | 0 | 1 | 0
  Causality: possibly related | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Causality: probably related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Causality: definetly related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severity: mild | 3 | 0 | 2 | 3 | 3 | 1 | 1 | 0
  Severity: moderate | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Severity: severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severity: life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severity: death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Reported Skin Reactions
Description: Local tolerability reactions, such as Erythema, swelling, pruritus, burning, blistering and urticaria, discolouration and dryness (Investigator's assessment 0-3 none/mild/moderate/severe).
Time Frame: Day 1 to Day 7.
Population: Full analysis set (FAS) consisted of all enrolled participants who received IMP.
Measure: Number; unit: participants
Groups:
- Part B, Cohort 1: 13 mg/cm2 GZ21T were applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 12 g cream.
- Part B, Cohort 2: 8 mg/cm2 GZ21T were applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 7 g cream.
- Part B, Cohort 3: 6,5 mg/cm2 GZ21T were applied to 900 cm2 of the skin, corresponding to approximately 5% BSA and 6 g cream.
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo | Part B, Cohort 1 | Part B, Cohort 2 | Part B, Cohort 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 3 | 3 | 3
participants
  Any erythema | 2 | 0 | 0 | 4 | 2 | 0 | 0 | 0
  Any swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any pruritus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any burning | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Any blistering | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any urticaria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any discoloration | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any dryness | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants in Part A with clinically significant changes from baseline in vital signs (systolic, diastolic blood pressure and pulse)
Time Frame: Day 1 to Day 7.
Population: Full analysis set (FAS) consisted of all enrolled participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants
  Systolic blood pressure | 0 | 0 | 0 | 0 | 0
  Diastolic blood pressure | 0 | 0 | 0 | 0 | 0
  Pulse | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiograms (ECGs)
Description: Number of participants in Part A with clinically significant changes from baseline in ECG results (resting heart rate, PQ/PR, QRS, QT and QTcF).
Time Frame: Day 1 to Day 7.
Population: Full analysis set (FAS) consisted of all enrolled participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants
  Resting heart rate | 0 | 0 | 0 | 0 | 0
  PQ/PR | 0 | 0 | 0 | 0 | 0
  QRS | 0 | 0 | 0 | 0 | 0
  QT | 0 | 0 | 0 | 0 | 0
  QTcF | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Test Results (Haematology, Clinical Chemistry, Coagulation)
Description: Number of participants in Part A with clinically significant abnormal laboratory tests results (clinical chemistry, hematology and coagulation parameters).
Time Frame: Day 1 to Day 7.
Population: Full analysis set (FAS) consisted of all enrolled participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants
  Haematology | 0 | 0 | 0 | 0 | 0
  Clinical chemistry | 0 | 0 | 0 | 0 | 0
  Coagulation | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Findings.
Description: Number of participants in Part A with clinically significant changes from baseline in physical examination findings.
Time Frame: Day 1 to Day 7.
Population: Full analysis set (FAS) consisted of all enrolled participants who received IMP.
Measure: Number; unit: participants
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Amount of Cream Absorbed After Single Dose Applications.
Description: Cream absorption measured on a 4-point scale: "1= not absorbed"; "2= somewhat absorbed"; "3= mostly absorbed"; "4= completely absorbed".
  This outcome was prespecified to be assessed only for Part B.
Time Frame: 0-2 hours after IMP administration
Population: All participants in Part B.
Measure: Number; unit: participants
Arm/Group | Part B, Cohort 1 | Part B, Cohort 2 | Part B, Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
participants
  30 min post-dose. Score 1 - not absorbed | 0 | 0 | 0
  30 min postdose. Score 2 - somewhat absorbed | 3 | 3 | 2
  30 min postdose. Score 3 - mostly absorbed | 0 | 0 | 1
  30 min postdose. Score 4 - completely absorbed | 0 | 0 | 0
  1 hour post-dose. Score 1 - not absorbed | 0 | 0 | 0
  1 hour postdose. Score 2 - somewhat absorbed | 3 | 3 | 0
  1 hour postdose. Score 3 - mostly absorbed | 0 | 0 | 3
  1 hour postdose. Score 4 - completely absorbed | 0 | 0 | 0
  2 hours post-dose. Score 1 - not absorbed | 0 | 0 | 0
  2 hours postdose. Score 2 - somewhat absorbed | 3 | 3 | 0
  2 hours postdose. Score 3 - mostly absorbed | 0 | 0 | 3
  2 hours postdose. Score 4 - completely absorbed | 0 | 0 | 0

8. Secondary Outcome: Plasma Concentrations
Description: Plasma concentrations of GZ21T after single dose applications.
Time Frame: Day 1 to Day 7.
Reporting Status: Not Posted

9. Secondary Outcome: PK Parameters- AUCinf
Description: PK parameters after a single dose application (to be calculated if data permits): area under the plasma concentration curve from time 0 to infinity (AUCinf).
Time Frame: Day 1 to Day 7.
Reporting Status: Not Posted

10. Secondary Outcome: PK Parameters - AUClast
Description: PK parameters after a single dose application (to be calculated if data permits): AUC from time 0 to the last measurable concentration (AUClast).
Time Frame: Day 1 to Day 7.
Reporting Status: Not Posted

11. Secondary Outcome: PK Parameters - Cmax
Description: PK parameters after a single dose application (to be calculated if data permits): maximum plasma concentration (Cmax).
Time Frame: Day 1 to Day 7.
Reporting Status: Not Posted

12. Secondary Outcome: PK Parameters - Tmax
Description: PK parameters after a single dose application (to be calculated if data permits): time to Cmax (Tmax).
Time Frame: Day 1 to Day 7.
Reporting Status: Not Posted

13. Secondary Outcome: PK Parameters - T½
Description: PK parameters after a single dose application (to be calculated if data permits): terminal elimination half-life (T½).
Time Frame: Day 1 to Day 7.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs (including serious AEs [SAEs]) were collected from the start of IMP administration until the end-of-trial visit of each part, from day 1 to day 7.
Description: The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. AEs were assessed as not related, unlikely related, or possibly, probably or definitely related to the IMP.
Arm/Group | Part A, Cohort 1 | Part A, Cohort 2 | Part A, Cohort 3 | Part A, Cohort 4 | Part A: Placebo | Part B, Cohort 1 | Part B, Cohort 2 | Part B, Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6 | 0/8 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6 | 2/6 | 3/6 | 3/8 | 1/3 | 1/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Cohort 1 (N=6) | Part A, Cohort 2 (N=6) | Part A, Cohort 3 (N=6) | Part A, Cohort 4 (N=6) | Part A: Placebo (N=8) | Part B, Cohort 1 (N=3) | Part B, Cohort 2 (N=3) | Part B, Cohort 3 (N=3)
Catheter site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The event was assessed as moderate in intensity and as not related to treatment with the IMP (applied 16 days prior to symptom onset).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Cohort 1 (N=6) | Part A, Cohort 2 (N=6) | Part A, Cohort 3 (N=6) | Part A, Cohort 4 (N=6) | Part A: Placebo (N=8) | Part B, Cohort 1 (N=3) | Part B, Cohort 2 (N=3) | Part B, Cohort 3 (N=3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results from this trial may be submitted for publication at the discretion of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT06888362/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT06888362/SAP_001.pdf